CLINICAL TRIAL: NCT02207504
Title: A Phase 1 Study of Crizotinib in Combination With Enzalutamide in Metastatic Castration-resistant Prostate Cancer Before or After Progression on Docetaxel.
Brief Title: Crizotinib in Combination With Enzalutamide in Metastatic Castration-resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Astellas Pharma Inc (Industry); Pfizer (Industry)
Responsible Party: Principal Investigator, Christopher Sweeney, MBBS, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-230
Record Dates: First submitted 2014-07-30; First posted 2014-08-04 (Estimated); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Castration-resistant Prostate Cancer
Keywords: Castration-resistant Prostate Cancer
MeSH Terms: interventions — Crizotinib; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- crizotinib and enzalutamide (Experimental): A traditional 3+3 dose escalation scheme will be used to identify the recommended phase 2 dose (RP2D) of crizotinib when used in combination with standard fixed dose enzalutamide.
  * Crizotinib- given orally daily-28 day cycle
  * Enzalutamide- given orally daily-28 day cycle
  Interventions: Drug: Crizotinib; Drug: Enzalutamide

INTERVENTIONS:
Drug: Crizotinib — Crizotinib is an ATP-competitive small-molecule inhibitor of the ALK, c-Met/HGFR, RON, and ROS receptor tyrosine kinases.
  Other Names: Xalkori; PF-02341066
Drug: Enzalutamide — Enzalutamide is an androgen receptor signaling inhibitor.
  Other Names: XTANDI; MDV3100

SUMMARY:
This research study is comparing the combination of drugs Crizotinib and Enzalutamide as a possible treatment for metastatic castration-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
* A traditional 3+3 dose escalation scheme will be used to identify the recommended phase 2 dose (RP2D) of crizotinib when used in combination with standard fixed dose enzalutamide.
* Patients who fulfill eligibility criteria will be entered into the trial to receive crizotinib and enzalutamide.
* After the screening procedures confirm participation in the research study:

  * The participant will be given a study drug-dosing calendar for each treatment cycle. The investigators are looking for the highest dose of the combination of study drugs that can be administered safely without severe or unmanageable side effects in participants that have, not everyone who participates in this research study will receive the same dose of the study drug. The dose given will depend on the number of participants who have been enrolled in the study prior and how well the dose was tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory and diagnostic tests, such as MRIs and CT scans, required for eligibility must be documented from tests performed within 30 days prior to the date of registration.
* The patient has pathologically confirmed adenocarcinoma of the prostate
* The subject must have CRPC with castrate levels of serum testosterone less than 50 ng/dL.

  -- NOTE: Subjects must maintain a castrate state. If they have not had an orchiectomy must continue to receive LHRH or GnRH agonists unless intolerant.
* Evidence of metastatic disease by radiographic imaging (bone scan or other nodal or visceral lesions on CT or MRI)
* Prostate cancer progression since last prior therapy documented by PSA according to PCWG2 or radiographic progression according to modified RECIST criteria Version 1.1
* No limit on number or type of prior therapies

  * Prior treatment with docetaxel is permitted but not required
  * Prior treatment with ketoconazole, estrogens, abiraterone or novel antiandrogens allowed, including past enzalutamide
  * Require at least a 6 week withdrawal period from the last dose of bicalutamide, or nilutamide or 4 weeks from last flutamide or enzalutamide dose Must have a documented PSA rise after stopping the antiandrogen --- Will require a 2 week washout period from last dose of ketoconazole, chemotherapy, or radiation
* Prior radiation is allowed
* Age ≥18 years
* ECOG performance status <2 (See Appendix 1)
* Life expectancy of greater than 6 months
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥1,500/mcL
  * Hemoglobin ≥8 g/dL

    ---*Transfusions and erythropoietin supplementation permitted
  * Platelets ≥100,000/mcL
  * Total bilirubin within normal institutional limits (unless known Gilbert's syndrome)
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal or ≤5X if presence of liver metastases

    --- *For patients with documented bone metastases, AST can be > 2.5x ULN if the investigator can provide evidence of no underlying liver dysfunction and thus, it is likely that the AST is originating from bone source.
  * Creatinine clearance ≥30 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* Able to swallow the study drug as a whole tablet
* The effects of crizotinib and enzalutamide on the developing human fetus are unknown. For this reason and because investigational agents as well as other standard antiandrogen agents used in this trial may be teratogenic, men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of crizotinib administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Pathology consistent with small cell carcinoma of the prostate
* Prior treatment with c-Met inhibitors
* Participants who have received any other investigational systemic agents in the last 2 weeks.
* Persistent grade >1 (NCI CTCAE v4.0) AEs due to investigational drugs that were administered more than 14 days before study enrollment with the exception of alocepia.
* Participants with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction or seizures that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to crizotinib or enzalutamide.
* History of seizure or any condition that may predispose to seizure (e.g., prior cortical stroke or significant brain trauma, history of loss of consciousness or transient ischemic attack within 12 months of study entry).
* Concomitant medications that would lower seizure threshold
* Concomitant use of medications that may alter pharmacokinetics of crizotinib or enzalutamide. See section 5.5, but would exclude the use of strong CYP3A or CYP2C8 inhibitors, strong or moderate CYP3A inducers, CYP2C8, CYP3A4, CYP2C9 and CYP2C19 substrates with narrow therapeutic indice.

  -- Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as: http://medicine.iupui.edu/clinpharm/ddis/table.aspx
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

  * Clinically significant heart disease defined as:

    * Myocardial infarction within 6 months of Screening visit.
    * Uncontrolled angina within 3 months of Screening visit.
    * Congestive heart failure New York Heart Association (NYHA) class 3 or 4, or subjects with history of congestive heart failure NYHA class 3 or 4 in the past, or history of anthracycline or anthracenedione (mitoxantrone) treatment, unless a screening echocardiogram or multi-gated acquisition scan (MUGA) performed within three months of the Screening visit results in a left ventricular ejection fraction that is ≥45%.
    * History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsade de pointes).
    * Prolonged corrected QT interval by the Fridericia correction formula (QTcF) on the screening electrocardiogram (ECG) > 470 msec.
    * History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place.
    * Hypotension (systolic blood pressure <86 mmHg) or bradycardia with a heart rate of <50 beats per minute on the Screening ECG, unless pharmaceutically induced and thus reversible (i.e. beta blockers) or known, chronic asymptomatic baseline heart rate.
    * Uncontrolled hypertension as indicated by a resting systolic blood pressure >170 mmHg or diastolic blood pressure >105 mmHg at the Screening visit.
    * No medications known to prolong the QT interval as crizotinib may increase the risk for QT prolongation
  * Thrombosis or vascular ischemic events within the last six months, such as deep venous thrombosis, pulmonary embolism, transient ischemic attack, cerebral infarction, or myocardial infarction
* No medications known to prolong the QT interval as crizotinib may increase the risk for QT prolongation
* Pregnant women are excluded from this study because women do not get prostate cancer, as they have no prostate.
* No defined washout period from major or minor surgery is required but incisions must be fully healed.
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with crizotinib or enzalutamide. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-08; Primary Completion 2018-02-02 (Actual); Study Completion 2022-01-03 (Actual)

PRIMARY OUTCOMES:
Rate of dose limiting toxicity (DLT) | 28 Days
  Rate of dose limiting toxicity (DLT) in the first 28 days of study therapy by dose level when escalating doses of crizotinib are combined with enzalutamide and when appropriate a GnRH agonist.

SECONDARY OUTCOMES:
Pharmacokinetics profiles of crizotinib and enzalutamide when used in combination | C1D1, C2D1: baseline, 0.5, 1, 2, 4, 6, and 8 hours after dose; prior to dose on C1D2, C2D2, C1D15, C2D15 , C3D1
  Pharmacokinetic parameters will be determined using noncompartmental methods with WinNonLin version 5.2. Maximum blood concentration (Cmax) and time of maximum blood concentration (tmax) will be determined by visual inspection. The area under the blood concentration-time curve (linear trapezoidal rule) will be determined between 0-24 hours (AUC0-24)/. The mean (+/- STDEM) concentration-time profiles of both crizotinib and enzalutamide will be presented for each dose.
The number of patients who experience adverse events and laboratory abnormalities | 2 Years
  The tolerability of the combination as defined as toxicity that results in study drug discontinuation or dose reduction that would not have been mandated by the protocol such as a DLT

OTHER OUTCOMES:
Time to radiologic disease progression | 2 years
  Time to radiographic progression based on the Kaplan-Meier Method from study entry to documented disease progression.
Blood markers of bone turnover and changes in bone microenvironment | 2 years
  Change in serum and bone-specific alkaline phosphatase and change in serum C-terminal telopeptides (CTx)
Change in quantity and gene expression of CTCs | 2 years
  Assessment of DNA alterations through whole exome sequencing and RNA analysis to assess the ability to detect the AR-V7 transcriptional variant and individual markers of AR and MET signaling using PCR-based methods
Time to disease progression including PSA | 2 years
  Time to radiographic progression based on the Kaplan-Meier Method from study entry to documented disease progression but with PSA values at corresponding timepoints.
Progression-free survival | 2 years
  Time to progression free survival based on the Kaplan-Meier Method from study entry to documented disease progression.
Time to treatment failure | 2 yrs
  Time to treatment failure from adverse event or progression
PSA response in patients who remain on therapy at 12 weeks | 2 yrs
  PSA response; change in alkaline phosphatase, CTx, and CTCs will be summarized descriptively

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sweeney, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No